CLINICAL TRIAL: NCT06934447
Title: Study of BCMA/CD70 Targeted Chimeric Antigen Receptor T (CAR- T) Therapy for Refractory Childhood-oneset Systemic Lupus Erythematosus
Brief Title: Study of BCMA/CD70 CAR-T Therapy for Refractory cSLE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Principal Investigator, Mao Jianhua, Professor, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC088
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: CAR T Cell Therapy; Systemic Lupus Erythematosus; BCMA
Keywords: systemic lupus erythematosus; Chimeric antigen receptor (CAR) T-cell; BCMA
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: Treatment of pediatric patients with refractory systemic lupus erythematosus using BMCA/CD70-targeted CAR T cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T treatment group (Experimental): This trial was designed as an open, single-arm, multicenter, dose-increasing trial.
  Interventions: Biological: anti-BCMA/CD70-CAR-T cells

INTERVENTIONS:
Biological: anti-BCMA/CD70-CAR-T cells — Three dose groups (0.3×105/kg, 1×105/kg, 3×105/kg) were set up, starting from the low dose group climbing to explore the safe and effective dose.

SUMMARY:
This is an investigator-initiated trial aimed at assessing the safety and efficacy of anti-BCMA/CD70 CAR-T cells in the treatment of refractory systemic lupus erythematosus.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a severe autoimmune disease that can lead to extensive damage in multiple organs and systems, potentially leading to disability and even mortality. Children afflicted with SLE are particularly vulnerable to organ damage, notably affecting the kidneys, and tend to have a more severe and protracted course of the disease compared to adults.

Currently, the primary treatment for SLE relies on glucocorticoids and immunosuppressants to alleviate symptoms. However, due to the absence of a curative treatment, patients typically need to remain on medication indefinitely. In recent years, biological agents such as belimumab and rituximab have been introduced for the treatment of SLE, but these treatments cannot completely eliminate autoimmune B cells in the bone marrow, leading to unsatisfactory overall outcomes. Furthermore, discontinuing these drugs can lead to disease relapse, and there is still no cure for SLE, leaving patients facing the challenges of lifelong medication and an incurable disease. BCMA (B Cell Maturation Antigen) is a receptor primarily expressed on the surface of mature B lymphocytes and plasma cells, serving as a marker protein for B lymphocyte maturation. B-cell activating factor (BAFF) and a proliferation-inducing ligand (APRIL) are the main ligands of BCMA. They interact with BCMA to transmit cellular stimulatory signals, activating TRAF-dependent NF-κB and JNK pathways, thereby increasing the proliferation and survival rate of B cells. Importantly, BCMA is highly expressed in long-lived plasma cells,8 which do not express CD19. Therefore, BCMA can compensate for the targeting defect of CD19's insufficient expression in terminally differentiated plasma cells. CD70 is an immune costimulatory molecule for T and B cells, highly expressed on the surface of activated T cells. The CD70/CD27 pathway regulates immunity and tolerance through various mechanisms, including T-cell expansion and survival, costimulation of antigen presentation, germinal center formation, B-cell activation, and antibody production. It plays a crucial role in the differentiation of B cells into plasma cells. Blocking the CD27/CD70 pathway can inhibit the differentiation of memory B cells into plasma cells. Studies have found that CD70 is overexpressed in B cells of SLE patients compared to healthy individuals.

The purpose of this study is to assess the safety and efficacy of the BCMA/CD70 CAR-T cells in the treatment of refractory SLE.

ELIGIBILITY:
Inclusion Criteria:

1. Age:≥5 years old;
2. Diagnosed with SLE according to the 2019 EULAR/ACR SLE classification criteria；Still in moderate to severe disease activity despite ≥3M of high dose glucocorticoids(prednisone≥1mg/kg/d or other equivalent amount of other steriod ), hydroxychloroquine and at least 2 of the following treatments(cyclophosphamide, MMF, azathioprine, methotrexate, cyclosporin, tacrolimus, sirolimus, leflunomide, telitacicept, Beliumab, and rituximab); or Intolerant to standard treatments;
3. SLEDAI 2K score≥8 points;
4. The functions of important organs are as follows: Cardiac function: Left ventricular ejection fraction (LVEF) ≥55% with no obvious abnormality in electrocardiogram; Renal function: eGFR≥30ML/min/1.73m2；Liver function: Asparagus cochinchinensis transase (AST) and Alanine Aminotransferase (ALT)≤3.0 ULN, Total Bilirubin (TBIL) in serum ≤2.0×ULN; Lung function: No serious lung lesions, SpO2≥92%;
5. No prior CAR-T therapy; or recurrence or poor response after previous treatment with autologous or allogeneic CAR-T targeting CD19 (as assessed by the investigator).
6. Met the standards of leukapheresis or intravenous blood collection, No contraindication for cell collection;
7. Negative pregnancy test for female Subjects of childbearing age, agree to take effective contraceptive measures the first year after CAR-T infusion;
8. Participants or their guardians agrees to participate in the clinical trial and sign the informed consent form which indicating that he/she understands the purpose and procedure of the clinical trial and is willing to participate in the study.

Exclusion Criteria:

1. Central nervous system (CNS) disease: CNS neurolupus requires intervention within 60 days);
2. Severe acute nephritis: Patients who have accepted or was undergoing renal replacement therapy within 3 months prior to transfusion; Or in the investgator's opinion, patients who is likely to have significant kidney disease within 3 moths of the study which need high dose glucocorticoid (prednisone dose≥1mg/kg/day or equivalent amount of other steriod), cyclophosphamide, or MMF treatment;
3. Have a history of congenital heart disease or acute myocardial infarction within 6 months prior to screening; Or severe arrhythmias (including multisource frequent supraventricular tachycardia, ventricular tachycardia, etc.); Or combined with moderate to massive pericardial effusion, serious myocarditis, etc; Or patients with unstable vital signs who need hypertensive drugs；
4. Suffer from other diseases that require long-term use of glucocorticoid or high-dose of immunosuppressive agents;
5. Uncontrollable infection, or active infection that requires systemic treatment within 1 week prior to screening；
6. History of organ transplantation or hematopoietic stem cell transplantation, or ≥Grade 2 GVHD within 2 weeks prior to screening；
7. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer greater than the normal reference value range; Or hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA titer greater than the normal reference value range; Or positive for human immunodeficiency virus (HIV) antibodies; Or syphilis test positive; Or cytomegalovirus (CMV) DNA test positive;
8. Received live vaccine within 4 weeks before screening;
9. Tested positive in Blood pregnancy test；
10. Previous or concurrent malignancy；
11. Patients who participated in other clinical study within 1 months prior to enrollment; Any other conditions that the investigators deem it unsuitable for the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
The safety of BCMA/CD70 CAR-T cell therapy in patients with refractory SLE | 3 months
  Incidence and severity of AEs and SAEs,including changes in laboratory values, Electrocardiograph(ECG) and vital signs assessed by CommonTerminology Criteria for Adverse Events (CTCAE) v5.0.
The efficiency of CAR-T cell therapy in patients with refractory SLE | 6 months
  Number of patients with SRI-4 response:including SLEDAI-2K ≥ 4-Point improvement, PGA with no worsening (&lt;0.3-point increase), BILAG 2004 with no new A domain score and no more than 1 new B domain scores. Number of patients with DORIS: including SLEDAI-2K = 0 and a Physician's Global Assessment (PGA) < 0.5, irrespective of serology, with permitted use of antimalarials, low-dose glucocorticoids (GCs; prednisolone ≤ 5 mg/day), and/or stable immunosuppressives and biologics.

SECONDARY OUTCOMES:
Cellular kinetics | 6 months
  CAR transgene levels by quantitative polymerase chain reaction (qPCR) in peripheral blood.
Autoantibody detection | 24 months
  Autoantibody detection up after BCMA/CD70 CAR-T cells infusion.
Pharmacokinetic Outcome AUC | 3 months
  The area under the curve (AUC) at 28 days and 90 days post-infusion (AUC28d/90d)
Duration of disease response (DOR) | 24 months
  The time between the first investigator assessment of remission and the first investigator assessment of progression or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Mao, MD, Principal Investigator — Zhejiang University School of Medicine Children's Hospital
Locations (1):
- hildren's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mackensen A, Muller F, Mougiakakos D, Boltz S, Wilhelm A, Aigner M, Volkl S, Simon D, Kleyer A, Munoz L, Kretschmann S, Kharboutli S, Gary R, Reimann H, Rosler W, Uderhardt S, Bang H, Herrmann M, Ekici AB, Buettner C, Habenicht KM, Winkler TH, Kronke G, Schett G. Anti-CD19 CAR T cell therapy for refractory systemic lupus erythematosus. Nat Med. 2022 Oct;28(10):2124-2132. doi: 10.1038/s41591-022-02017-5. Epub 2022 Sep 15. PMID 36109639
- [Background] Charras A, Smith E, Hedrich CM. Systemic Lupus Erythematosus in Children and Young People. Curr Rheumatol Rep. 2021 Feb 10;23(3):20. doi: 10.1007/s11926-021-00985-0. PMID 33569643
- [Background] Accapezzato D, Caccavale R, Paroli MP, Gioia C, Nguyen BL, Spadea L, Paroli M. Advances in the Pathogenesis and Treatment of Systemic Lupus Erythematosus. Int J Mol Sci. 2023 Mar 31;24(7):6578. doi: 10.3390/ijms24076578. PMID 37047548
- [Background] Schett G, Muller F, Taubmann J, Mackensen A, Wang W, Furie RA, Gold R, Haghikia A, Merkel PA, Caricchio R, D'Agostino MA, Locatelli F, June CH, Mougiakakos D. Advancements and challenges in CAR T cell therapy in autoimmune diseases. Nat Rev Rheumatol. 2024 Sep;20(9):531-544. doi: 10.1038/s41584-024-01139-z. Epub 2024 Aug 6. PMID 39107407
- [Background] Winter O, Dame C, Jundt F, Hiepe F. Pathogenic long-lived plasma cells and their survival niches in autoimmunity, malignancy, and allergy. J Immunol. 2012 Dec 1;189(11):5105-11. doi: 10.4049/jimmunol.1202317. PMID 23169863
- [Background] Liu Q, Deng Y, Liu X, Zheng Y, Li Q, Cai G, Feng Z, Chen X. Transcriptomic analysis of B cells suggests that CD70 and LY9 may be novel features in patients with systemic lupus erythematosus. Heliyon. 2023 Apr 23;9(5):e15684. doi: 10.1016/j.heliyon.2023.e15684. eCollection 2023 May. PMID 37144201
- [Background] Wang W, He S, Zhang W, Zhang H, DeStefano VM, Wada M, Pinz K, Deener G, Shah D, Hagag N, Wang M, Hong M, Zeng R, Lan T, Ma Y, Li F, Liang Y, Guo Z, Zou C, Wang M, Ding L, Ma Y, Yuan Y. BCMA-CD19 compound CAR T cells for systemic lupus erythematosus: a phase 1 open-label clinical trial. Ann Rheum Dis. 2024 Sep 30;83(10):1304-1314. doi: 10.1136/ard-2024-225785. PMID 38777376
- See also: BCMA-CD19 compound CAR T cells for systemic lupus erythematosus: a phase 1 open-label clinical trial. — https://pubmed.ncbi.nlm.nih.gov/38777376/
- See also: Transcriptomic analysis of B cells suggests that CD70 and LY9 may be novel features in patients with systemic lupus erythematosus. — https://pubmed.ncbi.nlm.nih.gov/37144201/
- See also: Anti-CD19 CAR T cell therapy for refractory systemic lupus erythematosus. — https://pubmed.ncbi.nlm.nih.gov/36109639/
- See also: Systemic Lupus Erythematosus in Children and Young People. — https://pubmed.ncbi.nlm.nih.gov/33569643/
- See also: Advances in the Pathogenesis and Treatment of Systemic Lupus Erythematosus — https://pubmed.ncbi.nlm.nih.gov/37047548/
- See also: Pathogenic long-lived plasma cells and their survival niches in autoimmunity, malignancy, and allergy. — https://pubmed.ncbi.nlm.nih.gov/23169863/